CLINICAL TRIAL: NCT02052349
Title: A Phase I, Open-Label Study to Investigate the Regional Bioavailability of ABT-333 When Delivered to Different Sites Within the Gastrointestinal Tract in Healthy Subjects
Brief Title: Bioavailability of ABT-333 Within the Gastrointestinal Tract in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M14-108; 2013-003161-34 (EudraCT Number)
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Relative Bioavailability
Keywords: relative bioavailability; healthy volunteers
MeSH Terms: interventions — dasabuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1: ABT-333 (Experimental): A single centre, open-label, 4-treatment, 3-period, 4-sequence incomplete randomised, single dose crossover study in healthy subjects.
  Interventions: Drug: ABT-333

INTERVENTIONS:
Drug: ABT-333 — Dose of ABT-333

SUMMARY:
This open label, Phase 1 study is to investigate the relative bioavailability of ABT-333 when delivered within different sites of the gastrointestinal tract in 12 healthy subjects.

DETAILED DESCRIPTION:
Bioavailability of ABT-333 in different areas of the gut

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
2. Subjects must demonstrate their ability to swallow an empty size 000 capsule
3. Must be willing and able to communicate and participate in the whole study
4. Must provide written informed consent
5. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. History of any drug or alcohol abuse in the past 2 years or current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
3. Females of childbearing potential who are pregnant or lactating (female subjects must have a negative urine pregnancy test at screening and admission)
4. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic xrays and other medical exposures, exceeding 5 (micro sievert) mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
5. Positive hepatitis A virus immunoglobulin M (HAVIgM), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
6. Donation or loss of greater than 400 mL of blood within the previous 3 months
7. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol, hormone replacement therapy (HRT) and hormonal contraception) or herbal remedies in the 14 days before Investigational Medical Product (IMP) administration. Exceptions may apply on a case by case basis if considered not to interfere with the objectives of the study by both the Principal Investigator (or delegate) and sponsor's medical monitor
8. Acute diarrhoea or constipation in the 7 days before the predicted first study day. If screening occurs >7 days before the first study day, this criterion will be determined on first study day. Diarrhoea will be defined as the passage of liquid faeces and/or a stool frequency of greater than 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day
9. Presence of non-removable metal objects such as metal plates, screws, etc, in the abdominal region of the body (with the exception of sterilisation clips)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ABT-333 drug concentrations | Day 1 until 24 hours after single dose of ABT-333 for each period
  ABT-333 concentrations in blood

SECONDARY OUTCOMES:
Physical Exam | Day-1 until 24 hours after single dose of ABT-333 for each period
  To examine any change from Day-1 in the subject's physical presentation(body temperature, pulse, blood pressure).
Electrocardiograms (ECGs) | Day-1 until 3 hours after single dose of ABT-333 for each period
  The measure of any change in 12 lead electrocardiogram from Day-1
Safety Labs | Day-1 until 24 hours after single dose ABT-333 for each period
  Chemistry, Hematology, Urinalysis
Number of participants with Adverse Events | Screening until after 7 days after last dose of ABT-333
Relative bioavailability | Day-1 until 24 hours after single dose of ABT-333 for each period
  The measure of ABT-333 in different areas of the gastrointestinal tract

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cohen, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 118435, Nottingham, United Kingdom